CLINICAL TRIAL: NCT00168467
Title: The Effects of Ramipril on Clinical Symptoms in Patients With Peripheral Arterial Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baker Heart Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20/03
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Ramipril

INTERVENTIONS:
Drug: Ramipril

SUMMARY:
One important clinical challenge in older individuals is maintaining mobility in the absence of pain. Peripheral arterial disease affects up to 12% of adults over 50 and impairs quality of life due to intermittent claudication causing pain and limiting mobility.

Conventional therapies have only modest effect in improving symptoms. The investigators hypothesise that angiotensin converting enzyme inhibition (with ramipril), which causes arterial vasodilation, also improves clinical symptoms in patients with peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria:

* Ankle-brachial index of <0.9 at rest in at least one leg
* History of intermittent claudication (unilateral or bilateral) which was stable for 6 months
* Evidence of superficial femoral artery stenosis or occlusion on duplex scan
* Blood pressure <=160/90 mmHg
* Stable medication regimen for at least 6 months and not previously treated with ACE inhibitors

Exclusion Criteria:

* Limiting coronary artery disease
* Renal Failure
* History of hypertension
* History of type 2 diabetes mellitus

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40

PRIMARY OUTCOMES:
Time to onset of claudication
Total exercise time during a standard treadmill test
Walking ability measured using the standard Walking Impairment Questionnaire

SECONDARY OUTCOMES:
Leg Blood Flow using Duplex Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn A Kingwell, PhD, Principal Investigator — Baker Heart Research Institute
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Result] Ahimastos AA, Lawler A, Reid CM, Blombery PA, Kingwell BA. Brief communication: ramipril markedly improves walking ability in patients with peripheral arterial disease: a randomized trial. Ann Intern Med. 2006 May 2;144(9):660-4. doi: 10.7326/0003-4819-144-9-200605020-00009. PMID 16670135 (Retraction: PMID 26544086 Ann Intern Med. 2015 Dec 1;163(11):884)